CLINICAL TRIAL: NCT02825368
Title: Homeopathic Vaccine Randomized Controlled Trial
Brief Title: Homeopathic Vaccine Trial
Acronym: HVT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HVT-2016
Record Dates: First submitted 2016-06-24; First posted 2016-07-07 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Homeopathic vaccine group (Experimental): * Diphtheria (Diphtherinum®), pertussis (Pertussinum®), tetanus (Tetanotxicum®), measles (Morbilinum®) and mumps (Ourlianum®) nosodes.
  * Two sterile saline injections (0.5ml each, intramuscular and subcutaneous) as placebo.
  Interventions: Other: Diphtherinum®; Other: Pertussinum®; Other: Tetanotxicum®; Other: Morbilinum®; Other: Ourlianum®; Other: Sterile saline
- Conventional vaccine group (Active Comparator): * One intramuscular dose of Tdap (tetanus, diphtheria, acellular pertussis)
  * One subcutaneous dose of MMR (measles, mumps, rubella)
  * Sugar pellets as placebo.
  Interventions: Biological: MMR; Biological: Tdap; Other: Sugar pellets
- Control group (Placebo Comparator): * Sugar pellets oral dose
  * Two sterile saline injections (0.5 ml each, intramuscular and subcutaneous) as placebo
  Interventions: Other: Sterile saline; Other: Sugar pellets

INTERVENTIONS:
Biological: MMR — 0.5 mL, subcutaneous
  Arms: Conventional vaccine group
Biological: Tdap — 0.5 mL, intramuscular
  Arms: Conventional vaccine group
Other: Diphtherinum®
  Arms: Homeopathic vaccine group
Other: Pertussinum®
  Arms: Homeopathic vaccine group
Other: Tetanotxicum®
  Arms: Homeopathic vaccine group
Other: Morbilinum®
  Arms: Homeopathic vaccine group
Other: Ourlianum®
  Arms: Homeopathic vaccine group
Other: Sterile saline — 0.5 mL, intramuscular
  Arms: Control group; Homeopathic vaccine group
Other: Sugar pellets
  Arms: Control group; Conventional vaccine group

SUMMARY:
The purpose of the study is to compare the immunological response of homeopathic vaccines to placebo and to conventional vaccines in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 24 years
* Has received primary childhood DTaP and MMR vaccinations
* Available for a follow up visit (3 weeks after initial visit)

Exclusion Criteria:

* Received a live vaccine in the past 4 weeks
* Has had a serious allergic reaction to a previous vaccination
* Has allergies to one or more of the components of the vaccines to be used (Neomycin, egg protein)
* Has a history of encephalopathy within 7 days of receiving DTP/DTap
* Has received nosodes for Diphtheria, Tetanus, Pertussis, Measles and Mumps
* Has received an adult booster dose of conventional vaccines of diphtheria, pertussis, tetanus, mumps, and measles (Tdap or MMR)
* Has received immunosuppressive doses of steroids or anti-cancer drugs in the past 3 months
* Is pregnant or if there is a chance they could become pregnant during the next month
* Has a moderate to severe acute illness at the time of enrolment
* Has cancer, leukemia, HIV/AIDS, or any other serious immune health condition
* Has a history of Guillaume Barre Syndrome
* Has received blood transfusion, blood products, or immune globulin within the past year

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Antibody levels for diphtheria | 3 weeks
Antibody levels for pertussis | 3 weeks
Antibody levels for tetanus | 3 weeks
Antibody levels for mumps | 3 weeks
Antibody levels for measles | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada